CLINICAL TRIAL: NCT05459779
Title: Evaluation of a Robotic Assistance Module for Driving Electric Wheelchairs Allowing the Avoidance of Positive and Negative Obstacles on the Driving Safety of Patients With Neurological Disorders.
Brief Title: Evaluation of a Robotic Assistance Module Against Positive and Negative Obstacles for Driving Electric Wheelchair
Acronym: SWADAPT 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Collaborators: INSA Rennes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-A00690-43
Record Dates: First submitted 2022-07-01; First posted 2022-07-15 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Neurological Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Each patient included will test a wheelchair equipped with a collision avoidance assistance module in 2 conditions, assistance activated or not.
Who Masked: Participant
Masking Description: To minimize bias, this study will be randomized and conducted in single blind. The patient will not be aware of the activation or not of the assistance module placed on the electric wheelchair. Indeed, the investigative team will be in charge of the activation of the robotic module.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric wheelchair with activated assistance module (Experimental): This condition will be achieved in a standardized test circuit composed by 9 platforms of increasing difficulty. The same day, the patient will perform the circuit 4 times, including 2 with activated assistance, in a random order established upstream.
  Interventions: Device: Electric wheelchair with activated assistance module
- Electric wheelchair with assistance module not activated (Other): This condition will be achieved in a standardized test circuit composed by 9 platforms of increasing difficulty. The same day, the patient will perform the circuit 4 times, including 2 without activated assistance, in a random order established upstream.
  Interventions: Device: Electric wheelchair with assistance module not activated

INTERVENTIONS:
Device: Electric wheelchair with activated assistance module — This evaluation will be carried out in 1 standardized test circuit composed by 9 platforms of increasing difficulty. The same day, the patient will perform the circuit 4 times, including 2 with activated assistance.
  Arms: Electric wheelchair with activated assistance module
Device: Electric wheelchair with assistance module not activated — This evaluation will be carried out in 1 standardized test circuit composed by 9 platforms of increasing difficulty. The same day, the patient will perform the circuit 4 times, including 2 without activating assistance.
  Arms: Electric wheelchair with assistance module not activated

SUMMARY:
The device that is the subject of this investigation is a robotic assistance module for driving a semi-autonomous electric wheelchair. This module is designed to accessorize the electric wheelchair to improve the safety conditions when driving an electric wheelchair, which on the one hand reduces the accident rate of wheelchair and on the other hand and facilitates the access to the wheelchair to people who cannot claim it without the use of a safety device of this type. The robotic assistance module is programmed to detect positive and negative obstacles.

DETAILED DESCRIPTION:
The device that is the subject of this investigation is a robotic assistance module for driving a semi-autonomous electric wheelchair. This module is designed to accessorize the electric wheelchair to improve the safety conditions when driving an electric wheelchair, thus reducing the wheelchair accident rate on the one hand and facilitating access to the wheelchair to persons who can not claim it without the use of a safety device of this type. The robotic assistance module is program to detect positive and negative obstacles.

This study "SWADAPT3" follows "SWADAPT1" and "SWADAPT2" with patients with Neurological Disorders, Regular Drivers of Electric Wheelchairs, in the same conditions:

Each patient included tested a wheelchair equipped with a collision avoidance assistance module in 2 conditions, assistance activated or not. This evaluation was carried out in 3 standardized test circuits of increasing difficulty, one week apart. At each session, the patient performed the circuit 6 times, including 3 with activated assistance, in a random order established upstream.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18,
* Having read the information note and freely consented to participate in the study,
* Suffering from neurological disorders such as cerebro-lesion or neuro-degeneration,
* Having benefited from an electric wheelchair prescription and/or learning to drive,
* The physical measurements (weight, height) are compatible with the use of the electric wheelchair chosen for the development of the robotics assistance module.

Exclusion Criteria:

* Understanding difficulties preventing the realization of the protocol,
* Motor disorders of the upper limb requiring additional driving technical assistance,
* Patient who has expressed difficulties impacting their internal and/or external driving safety,
* Pregnant, parturient or breastfeeding women,
* A person deprived of liberty by a judicial or administrative decision, persons under psychiatric care or admitted to a health or social institution for purposes other than research,
* Minors,
* a person in an emergency situation, unable to express his prior consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Success rate | Day 1
  Pass rate across standard platforms. The platform has been divided into sectors. The crossing of the platform stops as soon as a failure occurs (swing or collision). The circuit is composed of 9 platforms divided into 91 sectors. At the end, the success rate corresponds to the numbers of sector past with success with and without activation of the assistance system.
  Score rate : 0-91

SECONDARY OUTCOMES:
NASA-Task Load Index | Day 1
  The cognitive load of tests under both conditions will be measured by the NASA-Task Load Index. It is in the form of six scales where the participant must assign a score between zero and one hundred to each of them, score indicating a growing level of intensity. Three dimensions relate to the demands imposed on the subject (mental, physical and temporal demands) and three to the interaction of a subject with the task (effort, frustration and performance), with and without activation of the assistance system.
Calculated task load Index | Day 1
  During the evaluation, physiological signals (cardiac frequency /electroencephalography/Electro dermal activity) will be measured by skin sensors. The signals will be used to calculate a task load Index. The score ranges between 0 and 5 with 5 being the most demanding. The score will be measured before and after each condition.
Spontaneous stress assessment | Day 1
  The spontaneous stress measured by Visual Analogic Scale, from 0 to 100. The 0 represents not stressed at all and 100 extremely stressed. The score will be measured before and after each condition.
Calculated Stress Index | Day 1
  During the evaluation, physiological signals (cardiac frequency /electroencephalography/Electro dermal activity) will be measured by skin sensors. The signals will be used to calculate a Stress Index. The score ranges between 0 and 100 with 100 being the most stressful. The score will be measured before and after each condition.
Ease of Use Questionnaire | Day 1
  The satisfaction of the use of the electric wheelchair under the conditions will be evaluated by the self-questionnaire Ease of Use Questionnaire. It measures the subjective usability of a product or service. It is a 28-item survey that examines four dimensions of usability: usefulness, ease of use, ease of learning, and satisfaction. The questionnaires were constructed as seven-point Likert rating scales. Users were asked to rate agreement with the statements, ranging from strongly disagree (1) to strongly agree (7). The score will be measured after each condition.
UTAUT (Unified theory of acceptance of technology) questionnaire | Day 1
  Questionnaire of acceptability / acceptance of the tool and its use by patients based on the Unified Theory of Acceptance and Use Technology (UTAUT). The score will be measured at the end of the evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, Doctor, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pole Saint-Hélier, Rennes, Brittany Region, France